CLINICAL TRIAL: NCT06984315
Title: Spinal Anesthesia Mitigates Systemic Inflammatory Response Compared to General Anesthesia in Total Knee Arthroplasty: A Retrospective Study
Brief Title: Effects of Anesthesia Type on Inflammatory Response
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ali Genc, Assistant professor, Tokat Gaziosmanpasa University
Other Study IDs: 25-MOBAEK-160
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Spinal Aneshtesia; General Anesthetic; Inflammation; Neutrophils; Total Knee Arthroplasty; White Blood Cells
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group S: Underwent total knee arthroplasty under spinal anesthesia
  Interventions: Other: The effects of the groups on perioperative inflammation changes were compared.
- Group G: Underwent total knee arthroplasty under general anesthesia
  Interventions: Other: The effects of the groups on perioperative inflammation changes were compared.

INTERVENTIONS:
Other: The effects of the groups on perioperative inflammation changes were compared. — Between January 2020 and April 2025, data from 849 patients who underwent total knee arthroplasty were retrospectively reviewed. Preoperative hemogram values were obtained during routine anesthesia clinic evaluation, typically one day prior to surgery. Postoperative hemogram samples were collected on the day of surgery (postoperative day 0), within 4 to 12 hours after the procedure. Blood parameters included neutrophil, lymphocyte, monocyte, and platelet counts. Based on these values, inflammatory indices such as the neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), systemic immune-inflammation index (SII), and systemic inflammatory response index (SIRI) were calculated.

SUMMARY:
In total knee arthroplasty, surgical and anesthetic procedures can lead to a significant increase in systemic inflammation. This procedure is frequently performed under either general or spinal anesthesia. However, studies investigating the effect of anesthesia type on systemic inflammation have shown conflicting results. The Systemic Inflammatory Response Index (SIRI) and the Systemic Immune-Inflammation Index (SII) provide important information about the extent of systemic inflammation. This study aimed to investigate the effects of general and spinal anesthesia on perioperative changes in SII and SIRI during total knee arthroplasty. Between January 2020 and April 2025, data from 849 patients who underwent total knee arthroplasty were retrospectively reviewed. Patients received either spinal anesthesia (Group S) or general anesthesia (Group G). The groups were compared in terms of changes in perioperative SII and SIRI (ΔSII and ΔSIRI), total opioid consumption, postoperative complications, and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years
* Patients with ASA physical status I or II
* Patients who have underwent total knee arthroplasty under general or spinal anesthesia

Exclusion Criteria:

* Patients with BMI ≥40 kg/m2
* Patients with ASA physical status ≥III
* Patients with severe cardiopulmonary or metabolic disorders, coagulation disorders or active infection
* Patients with known allergies or chronic steroid use
* Patients with incomplete laboratory data
* Patients who underwent revision total knee arthroplasty
* Patients who required intraoperative conversion from spinal to general anesthesia
* Patients with a history of major trauma and/or emergency surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between January 2020 and April 2025, data from 849 patients who underwent total knee arthroplasty were retrospectively reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 849 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Systemic immune inflammation index (SII) and systemic inflammatory response index (SIRI) | Preoperative hemogram values were obtained during routine anesthesia clinic evaluation, typically one day prior to surgery. Postoperative hemogram samples were collected on the day of surgery (postoperative day 0), within 4 to 12 hours after the procedur
  SII = neutrophil X platelet / lymphocyte count and the SIRI = neutrophil X monocyte / lymphocyte count

SECONDARY OUTCOMES:
Neutrophil lymphocyte ratio (NLR) and platelet lymphocyte ratio (PLR) | Preoperative hemogram values were obtained during routine anesthesia clinic evaluation, typically one day prior to surgery. Postoperative hemogram samples were collected on the day of surgery (postoperative day 0), within 4 to 12 hours after the procedur
  NLR = neutrophil / lymphocyte and PLR= platelet / lymphocyte
Total amount of opioids consumed postoperatively | Total amount of opioids requirement within the first 24 postoperative hours
  Total opioid consumption was calculated by converting all opioid doses to morphine milligram equivalents

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data used to support the findings of this study can be obtained from the corresponding author on request.
Supporting Information: SAP